CLINICAL TRIAL: NCT00788138
Title: Effects of Vitamin D Supplementation on Lung Function in an Acute Pulmonary Exacerbation of Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Vin Tangpricha, Emory University School of Medicine
Organization: Atlanta VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Inpatient Vitamin D in CF
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Vitamin D; Anti-microbial peptides
MeSH Terms: conditions — Cystic Fibrosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Vitamin D3 250,000 PO Once
  Interventions: Dietary Supplement: Vitamin D3
- 2 (Placebo Comparator): Matching Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 250,000 IU of vitamin D3
  Other Names: Cholecalciferol
  Arms: 1
Dietary Supplement: Placebo — Matching Placebo
  Arms: 2

SUMMARY:
Vitamin D insufficiency is common in patients with cystic fibrosis. The investigators study will examine a large dose of vitamin D given to patients who have cystic fibrosis and are admitted to the hospital for a pulmonary exacerbation to determine whether vitamin D can improve clinical outcomes and whether the dose given is correct. The investigators hypothesis is that vitamin D therapy will improve production of anti-microbial peptides and will increase bacterial killing of microorganisms.

DETAILED DESCRIPTION:
Vitamin D insufficiency is common in CF patients. Treatment of vitamin D insufficiency in CF patients requires large doses of vitamin D. Adequate vitamin D status in CF is important for skeletal health and the prevention of osteoporosis. In addition to skeletal benefits of vitamin D, recent evidence has demonstrated that vitamin D plays an important role in the regulation of the immune system by increasing anti-microbial peptides in the lung and other barrier sites. Whether improving vitamin D status in CF patients would enhance the immune system has not yet been explored in a clinical study. This would have significant clinical impact in CF care since vitamin D status remains undertreated, especially in the setting of infection. The hypothesis of this proposal is that rapid correction of vitamin D insufficiency will result in improved innate immunity by increasing production of anti-microbial peptides resulting in more effective killing of bacteria. To address our hypothesis, the following two aims are proposed: 1) To evaluate the effect of rapid correction of vitamin D insufficiency as an adjunctive therapy on production of anti-microbial peptides in acute respiratory exacerbation in CF patients 2) To determine the effect of vitamin D treatment on bacterial killing in acute respiratory exacerbation in CF patients and to correlate with free LL-37 levels in sputum. The long term objective of this proposal and of our research group is to study the role of nutrition including vitamin D to improve the immune system in the setting of infection in CF.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria

* Study subjects must be patients diagnosed with cystic fibrosis and seen at the Emory University Cystic Fibrosis Center who are admitted to Emory University Hospital for an acute pulmonary exacerbation of cystic fibrosis as determined by their primary cystic fibrosis physician or emergency room physician.
* Study subjects must agree to participate in the study and provide written informed consent.
* Histology: Not applicable.
* Site: Emory University Hospital.
* Stage of Disease: Admission to Emory University Hospital for an acute pulmonary exacerbation of cystic fibrosis as determined by their primary CF physician based on symptoms and clinical evaluation.
* Age: Study subjects must be > 18 years old.
* Performance Status: Study subjects will be adult cystic fibrosis patients admitted to the hospital for an acute pulmonary exacerbation who are able to tolerate oral medication and to provide written informed consent.
* Informed Consent Requirement: All study subjects must agree to participate in the study and provide written informed consent, which will be written in English. An additional consent form will be provided to subjects who agree to long term storage of their blood, sputum, saliva, and exhaled breath for future use by investigators of this study.

Exclusion Criteria:

* Age < 18 years old.
* Inability to tolerate oral medications in the first 48 hours of admission.
* Prior other diseases: Patients with prior disorders potentially affecting vitamin D levels and metabolism of calcium and phosphate will be excluded. We will exclude patient with any known disorders of the endocrine system affecting vitamin D metabolism including: Hyperparathyroidism, known history of nephrolithiasis, any documented malignances, and advanced renal disease.
* Infection: Not applicable.
* Hematologic values that preclude entry into the study including serum creatinine > 1.5 mg/dL, to assist with exclusion of patients with renal disease, baseline serum 25-hydroxyvitamin D levels >80 ng/mL, and baseline calcium level > 10.5 mg/dL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Vitamin D status measured by serum 25-hydroxyvitamin D | 3 months
Antimicrobial peptide levels of LL-37, an endogenous anti-microbial peptide in humans | 3 months

SECONDARY OUTCOMES:
Markers of pulmonary function measured by FEV1 % predicted | 3 months
Length of hospitalization measured in days | 3 months
Number of days on antibiotic therapy | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States